CLINICAL TRIAL: NCT03633864
Title: Fecal Microbiota Transplantation for Refractory IgA Nephropathy: a Prospective, Single-center, Cohort Study
Brief Title: Fecal Microbiota Transplantation for Refractory IgA Nephropathy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Shiren sun, MD, Professor, Air Force Military Medical University, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMT for IgAN
Record Dates: First submitted 2018-08-07; First posted 2018-08-16 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: IgA Nephropathy
Keywords: IgA nephropathy; fecal microbiota transplantation
MeSH Terms: conditions — Glomerulonephritis, IGA | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FMT treatment (Experimental): FMT treatment arm: Accept fecal microbiota transplantation without changing the ongoing treatment strategy.
  Interventions: Biological: Fecal microbiota transplantation

INTERVENTIONS:
Biological: Fecal microbiota transplantation — Fecal donors are selected according to the predefined criteria. Fecal microbiota suspension is prepared by using fresh feces from the selected fecal donors. Then, administration of 200 ml fecal microbiota suspension through a transendoscopic enteral tubing or retention enema.

SUMMARY:
IgA nephropathy (IgAN) is one of the most common glomerular diseases worldwide. Current treatments for IgAN are limited by their relatively insufficient efficacy and severe adverse events. Previous studies suggested that the disorder of intestinal flora may play an important role in the pathogenesis and prognosis of IgAN. Fecal microbiota transplantation (FMT) have been proved to be effective on rebuilding the intestinal microecological balance. However, there is no evidence for the safety and efficacy of FMT in IgAN. Therefore, investigators perform a prospective cohort study to evaluate the safety and efficacy of FMT in IgAN patients who did not response to the conventional treatment and did not want to aggravate immunosuppressive treatments or IgAN patients who did not response to immunosuppressive treatments.

ELIGIBILITY:
Inclusion Criteria:

* Adult, age: 18-65 years old.
* Pathological diagnosis with IgAN, eGFR：20-120 mL/min/1.73 m2.
* The 24-hour urinary protein was still greater than 1g after 3-6 months of treatment of ACEI/ARB
* Recurrence of IgAN after glucocorticoid and (or)immunosuppressant decrement and the 24-hour urinary protein was greater than 1g.
* Not suitable for the administration of glucocorticoid and (or) immunosuppressive agents because of side effects.
* Women of child-bearing age with negative urine pregnancy test have no pregnancy plan for the next 18 months and take effective contraceptive measures.
* Agree to participate in this clinical trial

Exclusion Criteria:

* Malignant tumors and other diseases with expected survival time <3 months.
* Severe cardiovascular and cerebrovascular diseases and pulmonary dysfunction.
* Other immune system diseases.
* Diabetes
* Inflammatory bowel disease（IBD）
* Clostridium difficile infection
* Gastrointestinal tumor
* Active gastrointestinal bleeding
* Acute and chronic gastroenteritis
* Have received or are receiving FMT treatment.
* HIV
* Psychosis AND dysgnosia
* Contraindication of colonoscopy and enema
* Alcohol/drug abuse
* Other conditions that the researchers thought were not appropriate for the group.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-11-22 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Change of Urinary protein | one time per week up to 8 weeks
  24 hours urinary protein quantity

SECONDARY OUTCOMES:
Change of Serum creatinine | one time per week up to 8 weeks
  Concentration of serum creatinine
Change of eGFR | one time per week up to 8 weeks
  eGFR
Change of Hematuria | one time per week up to 8 weeks
  Hematuria
Change of Blood pressure | one time per week up to 8 weeks
  Blood pressure
Change of Serum IgA1 | one time per week up to 8 weeks
  Serum IgA1
Change of Fecal microbiota | one time per week up to 8 weeks
  Fecal microbiota
Adverse events associated with FMT | one time per week up to 8 weeks
  Adverse events associated with FMT

CONTACTS AND LOCATIONS:
Overall Officials: Shiren Sun, M.D., Principal Investigator — Xijing Hospital, the Fourth Military Medical University
Locations (1):
- Xijing Hospital of Nephrology, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided